CLINICAL TRIAL: NCT05832086
Title: Intermittent Fasting Using a Fasting-Mimicking Diet to Improve Prostate Cancer Control and Metabolic Outcomes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stephen Freedland (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Stephen Freedland, Director, Center for Integrated Research in Cancer and Lifestyle; Co-Director, Cancer Genetics and Prevention Program; Professor, Surger, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-02-FREEDLAND-FAST-PRO; 1R01CA280081-01 (NIH)
Record Dates: First submitted 2023-04-03; First posted 2023-04-27 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Prostate Adenocarcinoma
Keywords: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting Mimicking Diet (Experimental): Intermittent fasting using a fasting mimicking diet
  Interventions: Behavioral: Fasting Mimicking Diet (FMD)
- Standard Anti-Cancer Diet (Placebo Comparator): Standard Anti-Cancer Diet
  Interventions: Behavioral: Standard Anti-Cancer Diet

INTERVENTIONS:
Behavioral: Fasting Mimicking Diet (FMD) — Consume the FMD (Xentigen, L-Nutra, Los Angeles, CA) for 5 days every monthly cycle for 6 cycles total in 6 months.
  Arms: Fasting Mimicking Diet
Behavioral: Standard Anti-Cancer Diet — Will receive standard of care diet and exercise recommendations from the study dietitian. The diet advice will be consistent with the American Cancer Society for cancer survivors and exercise recommendation of a goal of 150 minutes/week of cardiovascular exercise and weight resistance training at least twice a week.
  Arms: Standard Anti-Cancer Diet

SUMMARY:
This is a Phase 2, randomized two-armed, multi-site study of 138 patients with metastatic castrate sensitive prostate adenocarcinoma. Patients will be randomized 1:1 to receive the fasting mimicking diet, or usual diet. All patients will receive standard of care treatment for their prostate cancer. The fasting mimicking diet will be consumed for 5 days per month for a total of 6 months and will be monitored by trained research dietitians.

This study aims to examine the effects of a fasting mimicking diet (5 days per month eating L-Nutra products only for 6 months) vs. usual diet on response to cancer treatment of metastatic castrate sensitive prostate adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castrate sensitive prostate adenocarcinoma (Adenocarcinoma prostate histologically confirmed by biopsy AND Metastatic disease confirmed biopsy, or MRI scan)
* Men receiving or planning to start first-line intensified ADT (within 30 days of registration) with abiraterone, apalutamide, enzalutamide, or darolutamide with or without current or prior chemotherapy
* Reads, writes, and understands English or Spanish and has telephone access for remote contact with the study dietitian.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Allergies to any ingredients listed on the Xentigen Ingredient List
* Men with diabetes who are not on stable doses of antihyperglycemic medication for at least 6 months and without physician consent that they may safely hold antihyperglycemic medication during the 5 days of FMD
* Regularly practicing a fasting diet that in the opinion of the study physician would impact study participation
* Significant co-morbidities (i.e., cardiac, pulmonary, liver disease, ongoing alcohol/drug abuse) that in the opinion of the study physician would preclude enrollment in this study.
* Body Mass Index (BMI) <20kg/m2
* Men actively trying to lose weight OR on weight loss medications (including but not limited to Contrave, Saxenda, Xenical) or planning to receive weight loss surgery in the next six months
* Self-reported weight loss ≥ 10% in the last 6 months

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Response to cancer treatment | 6 Month visit
  Will be measured by the proportion of patients who achieved PSA nadir ≤0.2 ng/dL at any time point within the 6-month study and absolute PSA nadir.

SECONDARY OUTCOMES:
Castration resistance 1 | 6 Month visit
  will be measured by Testosterone (ng/dl)
Castration resistance 2 | 6 Month visit
  will be measured by PSA levels (ng/mL)
Metabolic Toxicity 1 | Change from Baseline to 6 Month visit
  Will be measured by the changes in HbA1c
Metabolic Toxicity 2 | Change from Baseline to 6 Month visit
  Will be measured by the changes in waist circumference
Metabolic Toxicity 3 | Change from Baseline to 6 Month visit
  Will be measured by the changes in fat mass (assessed via bioelectrical expedience)
Metabolic Toxicity 4 | Change from Baseline to 6 Month visit
  Will be measured by the changes in body weight
Self-reported overall well-being | Change from Baseline to 6 Month visit
  will be measured in changes in the scores calculated from the Medical Outcomes Study Short Form Health Survey (SF-12) questionnaire. Scores can range from 12-56 with a higher score indicating a better outcome.
Self-reported energy levels | Change from Baseline to 6 Month visit
  will be measured in changes in the scores calculated from the Godin leisure-time physical activity questionnaire. Scores can range from 0 and above, with a higher score indicating a better physical activity outcome.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Beckman Research Institute of the City of Hope, Duarte, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No